CLINICAL TRIAL: NCT06195839
Title: Building Engagement Using Financial Incentives Trial - Hypertension
Acronym: BENEFIT-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020-1600-BENH
Record Dates: First submitted 2023-12-20; First posted 2024-01-08 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Health Behavior; Healthcare Patient Acceptance; Patient Engagement; Adherence, Patient
Keywords: preventive healthcare; patient financial incentives; federally qualified health center (FQHC); remote patient monitoring (RPM); health services
MeSH Terms: conditions — Hypertension; Health Behavior; Patient Acceptance of Health Care; Patient Participation; Patient Compliance | interventions — Remote Patient Monitoring

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Financial Incentives for BP monitoring (Experimental): * instructions for participating in a 2-month remote patient monitoring program
  * home blood pressure monitor and associated smartphone app, which includes a module for logging medication-taking
  * wrist-worn sensor and associated smartphone app
  * weekly adherence feedback to home blood pressure monitoring
  * immediate financial incentives for home blood pressure monitoring distributed weekly
  Interventions: Behavioral: Remote Patient Monitoring; Behavioral: Self-monitoring of hypertension-related factors; Behavioral: Immediate financial incentives
- Delayed Financial Incentives for BP monitoring (Active Comparator): * instructions for participating in a 2-month remote patient monitoring program
  * home blood pressure monitor and associated smartphone app, which includes a module for logging medication-taking
  * wrist-worn sensor and associated smartphone app
  * weekly adherence feedback to home blood pressure monitoring
  * delayed financial incentives for home blood pressure monitoring distributed at the end of the study
  Interventions: Behavioral: Remote Patient Monitoring; Behavioral: Self-monitoring of hypertension-related factors; Behavioral: Delayed financial incentives

INTERVENTIONS:
Behavioral: Remote Patient Monitoring — Participants will be given a home blood pressure machine and instructed to take their blood pressure twice/day (once in the morning and once at night) for the duration of the 2-month study. Blood pressure values will be immediately available in their patient-facing portal accessible via smartphone app, and patients will receive weekly feedback reports on their adherence to the home blood pressure monitoring protocol. Patients' blood pressure values will also be accessible to their clinical care team via an administrator portal, which will alert clinicians of any values above or below pre-specified clinical thresholds.
Behavioral: Self-monitoring of hypertension-related factors — As part of self-monitoring of hypertension-related factors, the blood pressure monitoring patient-facing app will also prompt patients daily to report whether or not they took their blood pressure medication. in addition, participants will be provided with a wrist-worn sensor and instructed to wear it at night to track their sleep activity. Data on sleep activity will be available to patients through a separate patient-facing app accessible on their smartphone.
Behavioral: Immediate financial incentives — Weekly financial incentives for measuring their blood pressure as instructed (up to $25/week: $5/day for up to 5 days/week)
  Arms: Immediate Financial Incentives for BP monitoring
Behavioral: Delayed financial incentives — Financial incentives for measuring their blood pressure as instructed in one payment at the end of the study (up to $25/week: $5/day for up to 5 days/week)
  Arms: Delayed Financial Incentives for BP monitoring

SUMMARY:
The goal of this pilot clinical trial is to determine feasibility and explore whether immediate versus delayed patient financial incentives improve patient engagement with self-monitoring of blood pressure in patients with uncontrolled hypertension at Louisiana federally qualified health centers (FQHCs). The main questions it aims to answer are:

* Do patients randomized to receive financial incentives on a weekly basis during the study (immediate) have better adherence to blood pressure self-monitoring compared to patients randomized to receive financial incentives at the end of the study (delayed)?
* Do patients randomized to immediate financial incentives have better blood pressure control compared to patients randomized to delayed incentives?

Participants will:

* attend a baseline visit to measure blood pressure, respond to a baseline survey, and receive remote patient monitoring devices and instructions to take home with them (home blood pressure monitor, wrist-worn sensor to track sleep activity, and associated apps)
* receive a random allocation to one of two groups: control condition (receive cash incentives at the end of the study for measuring blood pressure as instructed) or intervention condition (receive weekly cash incentives throughout the study for measuring blood pressure as instructed)
* use remote patient monitoring devices during a two month study period, receive weekly reports on adherence to blood pressure monitoring, and receive weekly financial incentives (intervention condition only)
* attend one follow-up visit at 2 months to measure their blood pressure, complete a follow-up survey, return the remote patient monitoring devices, and receive financial incentives for blood pressure monitoring (control condition only)

Researchers will compare the immediate and delayed incentive groups to see if there are differences in blood pressure monitoring adherence rates and blood pressure control.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years
* receive care at a participating FQHC
* taking blood pressure medication
* uncontrolled blood pressure at most recent clinic visit (systolic blood pressure ≥130 mm Hg or diastolic blood pressure ≥80 mm Hg)
* ability to understand and speak English
* able to access a smartphone

Exclusion Criteria:

* currently participating in another clinical trial or research study on blood pressure, medication-taking, or sleep
* unable or unwilling to give informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Between-group difference in weekly adherence to blood pressure monitoring | 8 weeks
  Weekly adherence to blood pressure monitoring will be defined as the number of days that the participant used the home blood pressure monitor at least once, captured in the blood pressure monitoring app usage data.

SECONDARY OUTCOMES:
Between-group mean difference in change in systolic blood pressure | 8 weeks
  Blood pressure will be measured at baseline and 8-week follow-up by a certified Clinical Research Coordinator using the average of three seated blood pressure measurements and in accordance with American Heart Association (AHA) guidelines.
Between-group mean difference in change in diastolic blood pressure | 8 weeks
  Blood pressure will be measured at baseline and 8-week follow-up by a certified Clinical Research Coordinator using the average of three seated blood pressure measurements and in accordance with American Heart Association (AHA) guidelines.
Between-group difference in the proportion with blood pressure control (<130/80 mm Hg) | 8 weeks
  Blood pressure will be measured at baseline and 8-week follow-up by a certified Clinical Research Coordinator using the average of three seated blood pressure measurements and in accordance with American Heart Association (AHA) guidelines. Blood pressure control will be defined as systolic <130 mm Hg and diastolic <80 mm Hg.
Between-group difference in the proportion with systolic blood pressure control (<130 mm Hg) | 8 weeks
  Blood pressure will be measured at baseline and 8-week follow-up by a certified Clinical Research Coordinator using the average of three seated blood pressure measurements and in accordance with American Heart Association (AHA) guidelines. Systolic blood pressure control will be defined as systolic <130 mm Hg.

OTHER OUTCOMES:
Number of patient approached for recruitment | 3 months
  Number of patients with reachable phone numbers or approached in clinic
Number of patients assessed for eligibility | 3 months
  Number of patients who begin eligibility screener
Number of patients enrolled | 3 months
  Number of patients who consent and are randomized
Number of patients who receive intended treatment | 2 months
  Proportion of total possible financial incentive received

CONTACTS AND LOCATIONS:
Overall Officials: Marie Krousel-Wood, MD, MSPH, Principal Investigator — Tulane University
Locations (2):
- United States (2):
  - CommuniHealth Services, Bastrop, Louisiana
  - David Raines Community Health Center, Shreveport, Louisiana